CLINICAL TRIAL: NCT07227038
Title: Living Well With Advanced Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Lilly Foundation (Unknown)
Responsible Party: Principal Investigator, Ashley Davenport, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-24331; NCI-2025-08030 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-11-07; First posted 2025-11-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Advanced Breast Carcinoma; Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients complete a survey and a semi-structured interview on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study

SUMMARY:
This study evaluates the use of supportive care in patients with advanced breast cancer to better understand what has helped them, what has been hard, and what kind of help they still need.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess acceptability of current LWABC model. II. Conduct a comprehensive review of participants' medical history, treatment records, and demographic data.

III. Explore differences in survivorship care engagement across four distinct cohorts.

OUTLINE: This is an observational study.

Participants complete a survey and a semi-structured interview on study.

ELIGIBILITY:
Inclusion Criteria:

* * COHORT 1:

  * Diagnosis of stage 4 metastatic breast cancer within the past 5 years
  * Never been referred to the LWABC
  * Adults age ≥ 18 years

    * COHORT 2:
  * Diagnosis of stage 4 metastatic breast cancer within the past 5 years
  * Have cancelled an appointment with the LWABC
  * Adults age ≥ 18 years

    * COHORT 3:
  * Been seen in the Medical Oncology Clinic at Stephanie Spielman Comprehensive Breast Center (SSCBC) within the past 5 years
  * Completed an appointment with the LWABC
  * Adults age ≥ 18 years

    * COHORT 4:
  * Caregivers for ABC patients
  * Adults age ≥ 18 years

Exclusion Criteria:

* Patients who cannot provide own informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with advanced breast cancer and their caregivers recruited through Ohio State University Comprehensive Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of current LWABC (Living Well with Advanced Breast Cancer) model | Up to study completion, up to 1 day
  Will utilize a thematic inductive analysis approach to compare and contrast themes across cohorts. Survey items will be summarized by cohort. Means, standard deviations, medians and ranges will be calculated for continuous variables and frequency, percents and 95% confidence intervals will be calculated for categorical variables.
Participant medical history, treatment records, and demographic data | Up to study completion, up to 1 day
  Will utilize a thematic inductive analysis approach to compare and contrast themes across cohorts. Survey items including demographic information and disease characteristics will be summarized by cohort. Means, standard deviations, medians and ranges will be calculated for continuous variables and frequency, percents and 95% confidence intervals will be calculated for categorical variables.
Differences in survivorship care engagement across four distinct cohorts | Up to study completion, up to 1 day
  Will utilize a thematic inductive analysis approach to compare and contrast themes across cohorts. Themes will be compared across each cohort to identify survivorship care needs that will be translated into intervention components for the ABC survivorship program. Survey items will be summarized by cohort. Means, standard deviations, medians and ranges will be calculated for continuous variables and frequency, percents and 95% confidence intervals will be calculated for categorical variables.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley P Davenport, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States